CLINICAL TRIAL: NCT00385489
Title: Single Ascending Dose Study of the Safety, Tolerability, and Pharmacokinetics of LXR-623 Administered Orally to Healthy Japanese Male Subjects.
Brief Title: Study Evaluating LXR-623 in Healthy Japanese Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3201A1-102
Record Dates: First submitted 2006-10-05; First posted 2006-10-09 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-08

CONDITIONS: Healthy
MeSH Terms: interventions — 2-(2-chloro-4-fluorobenzyl)-3-(4-fluorophenyl)-7-(trifluoromethyl)-2H-indazole

INTERVENTIONS:
Drug: LXR-623

SUMMARY:
The purpose of this study is to evaluate the safety of LXR-623 in healthy Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, Japanese Males aged 20-45 years

Exclusion Criteria:

* A history or active presence of clinically important medical disease

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2006-08; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Toshima-ku, Tokyo, Japan